CLINICAL TRIAL: NCT04226248
Title: CHolinesterase Inhibitor to prEvent Falls in Parkinson's Disease: A Phase 3 Randomised, Double-blind Placebo-controlled Trial of Rivastigmine to Prevent Falls in Parkinson's Disease.
Brief Title: CHIEF-PD (CHolinesterase Inhibitor to prEvent Falls in Parkinson's Disease)
Acronym: CHIEF-PD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Bristol (Other)
Collaborators: Royal United Hospitals Bath NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Study 2018-2030
Record Dates: First submitted 2019-12-05; First posted 2020-01-13 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Parkinson; Rivastigmine; Falls; Cholinesterase Inhibitors; Phase III
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: A Phase III Randomised Controlled Trial of Rivastigmine versus Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Rivastigmine) (Active Comparator): Rivastigmine Transdermal Patches
  Interventions: Drug: Rivastigmine Transdermal System
- Placebo (Placebo Comparator): Placebo Matched Transdermal Patches
  Interventions: Other: Placebo Transdermal System

INTERVENTIONS:
Drug: Rivastigmine Transdermal System — Rivastigmine Trandermal Patches applied once a day for up to 12 months
  Arms: Active (Rivastigmine)
Other: Placebo Transdermal System — Placebo Trandermal Patches applied once a day for up to 12 months
  Arms: Placebo

SUMMARY:
Parkinson's disease is a common condition particularly affecting older people. Falls are a very frequent complication of the disease affecting 60% of people with Parkinson's every year. As the population ages, the number of people living with Parkinson's disease and the occurrence of complications will increase. The loss of the chemical dopamine in the brain causes walking in Parkinson's to become slower, unsteady and irregular. People with the condition are therefore at a very high risk of falling. To some extent, people can compensate for these changes by paying more attention to their walking. However, Parkinson's also diminishes memory and thinking ability. This decreases people's ability to pay attention to their walking, especially when doing something at the same time.

Cholinesterase inhibitor (ChEis) are drugs that are currently used to treat people with memory problems in Parkinson's. The effect of these drugs on falls in Parkinson's has been tested to show that treatment has the potential to almost halve the number of falls.

This trial aims to definitively determine whether cholinesterase inhibitors (ChEi), can prevent falls in Parkinson's and whether this treatment is cost effective. 600 participants with Parkinson's disease will be enrolled from hospitals throughout the UK. Participants will be randomly assigned to either receive the drug (ChEi) via a patch or receive a placebo (dummy) treatment via a patch.

Neither the researchers nor the participants will know which group they are in. Participants will take the medication for 12 months and record any falls that they experience in diaries. If successful, this treatment in Parkinson's disease, would tackle one of the most disabling complications of the disease and positive findings will provide robust evidence to change clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease.
* Modified Hoehn and Yahr stage 1-4 disease as determined at baseline visit.
* Have experienced a fall in the previous year.
* Able to walk ≥10m without aids or assistance.
* 18+ years of age.

Exclusion Criteria:

* Previous ChEi use in 12 months prior to enrolment.
* Hypersensitivity to rivastigmine
* Dementia diagnosed according to MDS criteria (6).
* Inability to attend or comply with treatment or follow-up scheduling.
* Non-English-speaking patients (cognitive tests performed in English).
* Falling ≥4x per day.
* Unwillingness to use an acceptable method of contraception for the duration of the trial if they are of childbearing potential.
* Pregnancy and/or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Fall rate | 12 months from the day the IMP is commenced
  Fall rate measured using monthly diaries and telephone calls prospectively

SECONDARY OUTCOMES:
Parkinson's Disease (PD) | 12 months
  MDS-UPDRS total score in the practically defined 'ON' state and each individual subscale (1-4)
Freezing of gait | 12 months
  New Freezing of Gait Questionnaire (NFOGQ)
Frailty | 12 months
  Frailty assessed by the SHARE-FI
Physical performance | 12 months
  Measured by the Short physical performance battery (SPPB)
Freezing of Gait Assessment | 12 months
  Gait speed measured with Freezing of Gait (turn test)
Gait Assessment | 12 months
  Gait speed measured with and without dual task
Cognition | 12 months
  Montreal Cognitive Assessment (MoCA)
Depression | 12 months
  Geriatric Depression Scale (GDS)
Fear of falling | 12 months
  Iconographical Fall Efficacy Scale (ICON-FES)
Dysphagia | 12 months
  Swallowing Disturbance Questionnaire (SDQ)
Participant health related quality of life | 0,1,3,6 9 and 12 months
  EuroQoL 5D-5L health status questionnaire (EQ-5D-5L)
Capability of older people | 12 months
  ICEpop CAPability measure for Older people (ICECAP-O)
Mortality (all cause and PD-related) | 12 months
  Office of National Statistics (ONS) data
Cost effectiveness by NHS resource use | 12 months
  NHS Hospital Episode Statistics (HES) data
Apathy | 12 months
  Starkstein Apathy Scale

CONTACTS AND LOCATIONS:
Overall Officials: Emily Henderson, PhD, Principal Investigator — University of Bristol
Locations (38):
- United Kingdom (38):
  - Barking, Havering and Redbridge University Hospitals NHS trust, Romford, Accepted
  - Manchester University NHS Foundation Trust, Manchester, England
  - Betsi Cadwaladr University Health Board, Bangor, Gwynedd
  - Norfolk and Norwich University Hospital, Norwich, Norfolk
  - Lothian Health Board NHS, Edinburgh, Scotland
  - NHS Forth Valley, Larbert, Scotland
  - Royal United Hospitals Bath NHS Foundation Trust, Bath, Somerset
  - NHS Grampian, Aberdeen
  - Barnsley Hospital NHS Foundation Trust, Barnsley
  - University Hospitals Dorset NHS Foundation Trust, Bournemouth
  - Princess of Wales Hospital (Cwm Taf Morgannwg University Health Board), Bridgend
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol
  - North Bristol NHS Trust, Bristol
  - Pennine Acute Hospitals NHS Trust, Bury
  - University Hospitals of Derby and Burton NHS Foundation Trust, Derby
  - NHS Tayside, Dundee
  - Gateshead Health NHS Foundation Trust, Gateshead
  - Gloucestershire Hospitals NHS Foundation Trust, Gloucester
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - University Hospitals of Leicester NHS Foundation Trust, Leicester
  - The Walton Centre NHS Foundation Trust, Liverpool
  - Imperial College Healthcare NHS Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - South Tees Hospitals NHS Foundation Trust, Middlesbrough
  - Northumbria Healthcare NHS Foundation Trust, Newcastle
  - Newcastle Hospitals NHS Foundation Trust, Newcastle
  - Aneurin Bevan University Health Board, Newport
  - Oxford University Hospitals, Oxford
  - North West Anglia NHS Foundation Trust, Peterborough
  - University Hospitals Plymouth NHS Trust, Plymouth
  - Lancashire Teaching Hospitals NHS Foundation Trust, Preston
  - Royal Berkshire NHS Foundation Trust, Reading
  - Salford Royal NHS Foundation Trust, Salford
  - North Tees and Hartlepool Hospitals NHS Foundation Trust, Stockton-on-Tees
  - Somerset NHS Foundation Trust, Taunton
  - Wrightington, Wigan and Leigh Teaching Hospitals NHS Foundation Trust, Wigan
  - Betsi Cadwaladr University Health Board, Wrexham
  - Yeovil District Hospital, Yeovil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Neumann S, Taylor J, Bamford A, Metcalfe C, Gaunt DM, Whone A, Steeds D, Emmett SR, Hollingworth W, Ben-Shlomo Y, Henderson EJ. Cholinesterase inhibitor to prevent falls in Parkinson's disease (CHIEF-PD) trial: a phase 3 randomised, double-blind placebo-controlled trial of rivastigmine to prevent falls in Parkinson's disease. BMC Neurol. 2021 Oct 29;21(1):422. doi: 10.1186/s12883-021-02430-2. PMID 34715821